CLINICAL TRIAL: NCT06664268
Title: Clinical and Ultrasound Assessment of Efficacy of Plasma Rich Fibrin (PRF) Injection and Fractional CO2 Laser in Treatment of Postburn Hypertrophic Scars: a Randomized Controlled Clinical Trial
Brief Title: Effect of PRF & Fractional CO2 Laser in Postburn Hypertrophic Scars
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Emad Ahmed, plastic & reconstructive surgery Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRF&Laser in Postburn Scars
Record Dates: First submitted 2024-10-17; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Hypertrophic Scars; Burn Scar Patients
Keywords: PRF; Fractional CO2 Laser; Postburn Hypertrophic Scars
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): fractional CO2 laser alone
  Interventions: Device: Fractional CO2 laser assisted PDT
- Group B (Active Comparator): PRF Injection and fractional CO2 laser
  Interventions: Biological: Plasma rich in growth factors (PRGF-Endoret); Device: Fractional CO2 laser assisted PDT

INTERVENTIONS:
Biological: Plasma rich in growth factors (PRGF-Endoret) — Plasma Rich Fibrin (PRF) is a newer modality in regenerative medicine derived from the patient's own blood. PRF does not use anticoagulants during processing, leading to a natural fibrin matrix that supports prolonged release of growth factors and cytokines .This matrix has been shown to enhance wound healing and improve scar texture and appearance .
  Arms: Group B
Device: Fractional CO2 laser assisted PDT — Fractional CO2 laser therapy is a well-established technique for scar treatment, including postburn scars. This technology utilizes laser energy to create microthermal zones in the skin, which stimulates collagen production and skin remodeling while minimizing damage to surrounding tissues .

SUMMARY:
Recent advancements in scar management include the use of Plasma Rich Fibrin (PRF) injections and fractional CO2 laser treatments. Both modalities are considered innovative approaches that offer promising outcomes in scar revision .

Plasma Rich Fibrin (PRF) is a newer modality in regenerative medicine derived from the patient's own blood. Unlike platelet-rich plasma (PRP), PRF does not use anticoagulants during processing, leading to a natural fibrin matrix that supports prolonged release of growth factors and cytokines . This matrix has been shown to enhance wound healing and improve scar texture and appearance. Studies have demonstrated PRF's efficacy in treating various skin conditions, including acne scars and general skin rejuvenation, suggesting potential benefits for postburn scar management .

Fractional CO2 laser therapy is a well-established technique for scar treatment, including postburn scars. This technology utilizes laser energy to create microthermal zones in the skin, which stimulates collagen production and skin remodeling while minimizing damage to surrounding tissues . Clinical trials have validated the effectiveness of fractional CO2 lasers in reducing scar thickness and improving skin texture, making it a popular choice for scar revision .

DETAILED DESCRIPTION:
Postburn scars often result in significant functional and aesthetic challenges for plastic surgeons. These scars can cause physical limitations, psychological distress, and a decrease in quality of life. Traditional treatments, including topical therapies, silicone gel sheets, and surgical interventions, frequently fall short in providing optimal results, particularly for extensive or complex scars .

Recent advancements in scar management include the use of Plasma Rich Fibrin (PRF) injections and fractional CO2 laser treatments. Both modalities are considered innovative approaches that offer promising outcomes in scar revision .

Plasma Rich Fibrin (PRF) is a newer modality in regenerative medicine derived from the patient's own blood. Unlike platelet-rich plasma (PRP), PRF does not use anticoagulants during processing, leading to a natural fibrin matrix that supports prolonged release of growth factors and cytokines . This matrix has been shown to enhance wound healing and improve scar texture and appearance. Studies have demonstrated PRF's efficacy in treating various skin conditions, including acne scars and general skin rejuvenation, suggesting potential benefits for postburn scar management .

Fractional CO2 laser therapy is a well-established technique for scar treatment, including postburn scars. This technology utilizes laser energy to create microthermal zones in the skin, which stimulates collagen production and skin remodeling while minimizing damage to surrounding tissues . Clinical trials have validated the effectiveness of fractional CO2 lasers in reducing scar thickness and improving skin texture, making it a popular choice for scar revision .

Despite the individual benefits of PRF and fractional CO2 laser treatments, there is a lack of direct comparative studies assessing their relative efficacy in postburn scar management. Comparative research is essential to determine which treatment provides superior outcomes and to guide clinical decision-making .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 60 years
* Mature post burn scars (more than 6 months).
* Scar area does not exceed 5% of body surface area (TBSA).

Exclusion Criteria:

* Immature scars (less than 6 months).
* Large scar area (more than 5%of body surface area (TBSA).
* Previous scar treatment with other modalities.
* Keloid scars.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Assessment | 6 months
  1. Clinical Assessment:
  By Vancouver Scar Scale (VSS) which consists of four items:
  1. Pigmentation (0-2) Normal 0 Hypopigmentation 1 Hyperpigmentation 2
  2. Vascularity (0-3) Normal 0 Pink 1 Red 2 Purple 3
  3. Pliability (0-5) Normal 0 Supple 1 Yielding 2 Firm 3 Banding 4 Contracture 5
  4. Height (0-3) Normal (flat) 0 0-2 mm 1 2-5 mm 2 >5 mm 3 It has a score ranging from 0-13 , The VSS set a precedent for systematic scar assessment by collecting subjective assessments and using a semiquantitative approach. 0 (best) - 13 (worst)
Ultrasound Assessment | 6 months
  Ultrasound Assessment: to detect changes in hypertrophic scar thickness before, during, and after treatment By Measurement of
  * scar thickness in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Makboul, Professor, Study Director — Assiut University; Ahmed Ali, Assistant Proffesor, Study Director — Assiut University

REFERENCES:
- [Background] Arsiwala NZ, Inamadar AC, Adya KA. A Comparative Study to Assess the Efficacy of Fractional Carbon Dioxide Laser and Combination of Fractional Carbon Dioxide Laser with Topical Autologous Platelet-rich Plasma in Post-acne Atrophic Scars. J Cutan Aesthet Surg. 2020 Jan-Mar;13(1):11-17. doi: 10.4103/JCAS.JCAS_142_19. PMID 32655245
- [Background] Chen Y, Wei W, Li X. Clinical efficacy of CO2 fractional laser in treating post-burn hypertrophic scars in children: A meta-analysis: CO2 fractional laser in treating post-burn hypertrophic scars in children. Skin Res Technol. 2024 Feb;30(2):e13605. doi: 10.1111/srt.13605. PMID 38332516
- [Background] Godara S, Arora S, Dabas R, Arora G, Renganathan G, Choudhary R. A Comparative Study on the Efficacy of Fractional CO2 Laser and Fractional CO2 Laser with Autologous Platelet-Rich Plasma in Scars. Indian Dermatol Online J. 2020 Sep 19;11(6):930-936. doi: 10.4103/idoj.IDOJ_174_20. eCollection 2020 Nov-Dec. PMID 33344342
- [Background] Choi KJ, Williams EA, Pham CH, Collier ZJ, Dang J, Yenikomshian HA, Gillenwater TJ. Fractional CO2 laser treatment for burn scar improvement: A systematic review and meta-analysis. Burns. 2021 Mar;47(2):259-269. doi: 10.1016/j.burns.2020.10.026. Epub 2020 Nov 9. PMID 33288326
- [Background] Castro AB, Meschi N, Temmerman A, Pinto N, Lambrechts P, Teughels W, Quirynen M. Regenerative potential of leucocyte- and platelet-rich fibrin. Part A: intra-bony defects, furcation defects and periodontal plastic surgery. A systematic review and meta-analysis. J Clin Periodontol. 2017 Jan;44(1):67-82. doi: 10.1111/jcpe.12643. Epub 2016 Nov 24. PMID 27783851
- [Background] Manole CG, Soare C, Ceafalan LC, Voiculescu VM. Platelet-Rich Plasma in Dermatology: New Insights on the Cellular Mechanism of Skin Repair and Regeneration. Life (Basel). 2023 Dec 25;14(1):40. doi: 10.3390/life14010040. PMID 38255655
- [Background] Elver A, Caymaz MG. Novel approaches to the use of platelet-rich fibrin: A literature review. Saudi Dent J. 2023 Nov;35(7):797-802. doi: 10.1016/j.sdentj.2023.07.008. Epub 2023 Jul 10. No abstract available. PMID 38025602
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part I: technological concepts and evolution. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e37-44. doi: 10.1016/j.tripleo.2005.07.008. Epub 2006 Jan 19. PMID 16504849
- [Background] Tredget EE, Shupp JW, Schneider JC. Scar Management Following Burn Injury. J Burn Care Res. 2017 May/Jun;38(3):146-147. doi: 10.1097/BCR.0000000000000548. PMID 28338518
- [Background] Lang TC, Zhao R, Kim A, Wijewardena A, Vandervord J, Xue M, Jackson CJ. A Critical Update of the Assessment and Acute Management of Patients with Severe Burns. Adv Wound Care (New Rochelle). 2019 Dec 1;8(12):607-633. doi: 10.1089/wound.2019.0963. Epub 2019 Nov 6. PMID 31827977